CLINICAL TRIAL: NCT00971685
Title: Evaluation of Efficacy and Safety of Lenalidomide (Revlimid®) in Patients With POEMS Syndrome
Brief Title: The Treatment of Lenalidomide in Patients With POEMS Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Armando Santoro, MD, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2008-002
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: POEMS Syndrome
MeSH Terms: conditions — POEMS Syndrome | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide plus Dexamethasone (Experimental): RD regimen: Lenalidomide 25 mg/die for 21 days every month for 6 cycles, with once-weekly dexamethasone (40 mg).
  Interventions: Drug: Lenalidomide and dexamethasone

INTERVENTIONS:
Drug: Lenalidomide and dexamethasone — RD regimen: Lenalidomide 25 mg/die for 21 days every month for 6 cycles, with once-weekly dexamethasone (40 mg).

SUMMARY:
Lenalidomide is a immunomodulatory drug derived from thalidomide, without neurotoxicity. Lenalidomide blocks the increased secretion of interleukin-6, tumor necrosis factor alpha and vascular endothelial growth factor (VEGF). The association with dexamethasone increased Lenalidomide response rate.

More recently the efficacy of Lenalidomide has been reported in a patient with POEMS (POEMS:polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome with improvement of clinical condition and reduction of vascular endothelial growth factor (VEGF) and interleukin-6 (IL-6) level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of POEMS syndrome based on published diagnostic criteria

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical efficacy of Lenalidomide for 21 days every month for 6 cycles, with once-weekly dexamethasone (40 mg)) in patients with POEMS syndrome after 6 cycles. | one year

SECONDARY OUTCOMES:
Evaluation of the safety and the activity. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinco Humanitas, Rozzano, Milano, Italy